CLINICAL TRIAL: NCT05215067
Title: A Phase II Trial of AK104 in Combination With Docetaxel in Subjects With Advanced Non-Small Cell Lung Cancer and Progressive Disease After Platinum Doublet Chemotherapy and Treatment With One Prior Anti-PD-1/PD-L1 Monoclonal Antibody (mAb)
Brief Title: A Phase II Trial of AK104 in Advanced Non-Small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK104-215
Record Dates: First submitted 2022-01-18; First posted 2022-01-31 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Advanced Non-small Cell Lung Cancer
MeSH Terms: interventions — Docetaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK104 plus Docetaxel (Experimental): AK104 RP2D + Docetaxel 75mg/m^2 every 3 weeks until progressive disease or unacceptable toxicity.
  Interventions: Drug: AK104; Drug: Docetaxel

INTERVENTIONS:
Drug: AK104 — IV infusion,Specified dose on specified days
Drug: Docetaxel — IV infusion,Specified dose on specified days

SUMMARY:
Phase II open label, multicenter study to evaluate the efficacy and safety of AK104 (anti-PD-1 and CTLA-4 bispecific antibody) combined with Docetaxel in Advanced Non-Small Cell Lung Cancer whose disease has progressed after prior platinum doublet chemotherapy and anti-PD-1/PD-L1 monoclonal antibody

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 75 years old.
2. Have a life expectancy of at least 3 months.
3. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Has a histologically or cytologically confirmed diagnosis of locally advanced or metastatic NSCLC.
5. Has radiographic progression after prior platinum doublet chemotherapy and anti-PD-1/PD-L1 monoclonal antibody (mAb) administered.
6. No known epidermal growth factor receptor (EGFR) or anaplastic lymphoma kinase (ALK) mutations.
7. Has at least 1 measurable lesion per RECIST 1.1 assessed by investigator.
8. Has adequate organ function.

Exclusion Criteria:

1. Undergone major surgery within 30 days prior to the first dose of study treatment.
2. Active central nervous system (CNS) metastases.
3. History of active autoimmune disease that has required systemic treatment in the past 2 years (i.e.,corticosteroids or immunosuppressive drugs).
4. Active Hepatitis B or Hepatitis C.
5. Received previous immunotherapy, including immune checkpoint inhibitors, immune checkpoint agonists, immune cell therapy and other treatments targeting the mechanism of tumor immunity.
6. Has received treatment with docetaxel.
7. History of severe bleeding tendency or coagulation disorder.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 2 years

SECONDARY OUTCOMES:
Number of patients with Adverse Events (AEs) | Up to approximately 2 years
  Characterization of incidence, severity and abnormal clinically significant laboratory findings of AEs
Disease control rate (DCR) | Up to approximately 2 years
Duration of Response (DOR) | Up to approximately 2 years
Time to response (TTR) | Up to approximately 2 years
Progression free survival (PFS) | Up to approximately 2 years
Overall survival (OS) | Up to approximately 2 years
Pharmacokinetic Parameter Area Under the Plasma Concentration-Time Curve (AUC) Of AK104 | Up to approximately 2 years
Antidrug antibodies (ADA) of AK104 | Up to approximately 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Cancer Hospital, Nanjing, Jiangsu, China